CLINICAL TRIAL: NCT02957903
Title: Sensory Distribution of Lateral Femoral Cutaneous Nerve Block - A Randomized, Blinded, Paired Trial in Healthy Volunteers
Brief Title: Sensory Distribution of Lateral Femoral Cutaneous Nerve Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Naestved Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SM1-KHT-2016; 2016-002643-41 (EudraCT Number)
Record Dates: First submitted 2016-10-31; First posted 2016-11-08 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2016-10

CONDITIONS: Nerve Block; Anesthesia, Local; Pain, Postoperative; Anatomical Distribution
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): Injection around the lateral femoral cutaneous nerve:
  8 ml Ropivacaine 0.75 %.
  Interventions: Drug: Ropivacaine
- Treatment B (Placebo Comparator): Injection around the lateral femoral cutaneous nerve:
  8 ml isotonic Saline.
  Interventions: Drug: Isotonic Saline

INTERVENTIONS:
Drug: Ropivacaine — All 20 study participants will receive both treatment A and B in form of a nerve block injection around the lateral femoral cutaneous nerve. Treatment A and B will be randomized to be given in either right or left lower extremity. If the participant is randomized to receive treatment A in the right lower extremity, treatment B will be given in the left lower extremity, and vice versa. Each participant will thus constitute as their own control.
  Other Names: 8 ml Ropivacaine 0.75 %
  Arms: Treatment A
Drug: Isotonic Saline — All 20 study participants will receive both treatment A and B in form of a nerve block injection around the lateral femoral cutaneous nerve. Treatment A and B will be randomized to be given in either right or left lower extremity. If the participant is randomized to receive treatment A in the right lower extremity, treatment B will be given in the left lower extremity, and vice versa. Each participant will thus constitute as their own control.
  Other Names: 8 ml isotonic Saline
  Arms: Treatment B

SUMMARY:
The purpose of this study is to investigate and describe the anatomical distribution of the sensory outcome following LFCN block (LFCN = lateral femoral cutaneous nerve) in relation to the incisional lines after Total Hip Arthroplasty (THA). Furthermore, is the aim to examine whether there is a motorial outcome corresponding to the Femoral nerve. The trial will be conducted in healthy volunteers in a blinded, randomized paired study.

DETAILED DESCRIPTION:
Background:

Total hip arthroplasties may be associated with moderate to intense postoperative pain. It is essential that pain treatment, besides being analgesic, has a minimum of side effects, especially those opioid-related, in order to achieve low morbidity, high patient satisfaction and to encourage the functional rehabilitation.

Currently, there is no "gold standard" for pain treatment after THA, and there exists a large variety of treatment options. Some patients who have undergone THA, can be difficult to sufficiently treat with conventional analgesics without reaching additional morphine doses where side effects are unacceptable. It is therefore important to explore other treatment options, including nerve blockade.

Nerve blocks have previously been used after THA operations, but have been hampered by the fact, that the nerve blocks have an effect on the motorial nerve, inhibiting early mobilization and possibly increasing tendencies to fall when mobilized. LFCN is purely sensorial and can therefore relieve the patient of pain without influencing the early mobilization. In addition, the application of nerve blocks is very easy and virtually without complications.

In two previous trials, the investigators have studied the effect of LFCN blocks in pain treatment after THA. In the recent study, the LFCN block was applied in patients after THA, who still had visual analogue scale (VAS) mobilization pain > 40 mm when lifting their leg stretched. The LFCN block alleviated significantly the average pain at group level. Meanwhile 42% of patients in the study had no or limited effect of the block. The reason for this may be due to the fact, that LFCN block does not cover all types of pain after THA, but also the fact, that the nerve innervation area has individual differences in the anatomical distribution. It is therefore relevant to describe the anatomical distribution of a LFCN block in order to determine whether the variations in anatomy is a contributing factor of the high number of patients with no effect of the blockade.

An earlier study investigated the proportion of the incisional line associated with total hip arthroplasty that was covered by the LFCN block. However the study was not blinded or randomized, and the description of the anatomical distribution of the block was inadequate.

Methods:

Prior to applying the nerve block, the measurement methods are tested and baseline values are registered for each leg of each participant.

The effect of a nerve block in healthy individuals can be studied by a number of validated measurement techniques. These techniques consist of mapping the affected anatomical area with temperature discrimination test (cold sensation) by using alcohol soaked gauze and pin-prick test by using a Von Frey filament, and of a pain stimulation test with determination of the heat pain threshold (Heat Pain Detection Threshold, HPDT) and pain during tonic heat-stimulation of the skin (VAS tonic heat stimulation). The duration and distribution of the sensory block is thus evaluated by high precision.

It is furthermore important to investigate whether the nerve blockade affects N. Femoralis' motorial innervation by testing m.Quadriceps' motorial function.

Course of study:

1. Baseline values are measured.
2. An orthopedic surgeon draws two hypothetical incisional lines corresponding to the posterior and to the anterior-lateral access to the hip joint on each leg of each participant. The incisional lines will be drawn with UV paint only visible under UV light. No other than the person drawing the lines and the participant will see where the lines are drawn.
3. An ultrasound guided LFCN block is applied by a specialist in anesthesia. Each trial participant will get an injection of Ropivacaine (active ingredient) in one leg and an injection of isotonic NaCl (placebo) in the other leg. Neither trial participant, doctors or investigator will know which treatment the participant receives in which leg, that is the trial is blinded.
4. After the LFCN block is applied a line called "Line A" is drawn on each leg. Line A goes from trochanter major to the femoral lateral epicondyle and is extended cranial. A line 0A is drawn perpendicular on line A at the trochanter major point. 5 cm above line 0A, is line -1A drawn up to -3A, and 5 cm below line 0A is line 1A drawn, and so forth to line 15A is reached.
5. One hour after the nerve block is applied to the right leg, the motorial and sensorial tests will be carried out on each leg, and the outcome will be registered and documented with photography. The test will be carried out on the right leg and then on the left leg in following order:

   * Maximum isometric voluntary contraction
   * Temperature discrimination test (alcohol soaked gauze)
   * Pin-prick (Von Frey filament)
   * Photo documentation
   * Drawing of the incisional lines under UV-light
   * Photo documentation
   * Measurement of the incisional lines
   * Heat pain detection threshold test
   * Pain stimulation test.

The subjects will be monitored with blood pressure, pulse oximetry and ECG during the trial. The study extends for each participant from the introductory conversation to all testing is complete.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have given their written consent after understanding the content and limitations og the study.
* ASA 1-2.
* BMI ≥18 and ≤ 30

Exclusion Criteria:

* Participants who can not cooperate in the study.
* Participant who can not speak or understand danish.
* Allergies to the drugs used in the study.
* Alcohol consumption that exceeds 21 units per week.
* Drug abuse by the investigators judgement.
* Daily consumption of prescription required analgesic drugs within the last four weeks.
* Consumption of over the counter analgesic drugs within the last 48 hours.
* Neuromuscular defects, former surgery or trauma to the lower extremities.
* Diabetes mellitus.
* Pregnant women (women in the fertile age must have used safe contraception and test negative with a urine-HCG to be able to participate in the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Difference in the percentage coverage of the incision (posterior approach) assessed by cold sensation | 1 hour post-block
  Difference in the percentage coverage of the incision (posterior approach) between the side given Ropivacaine versus the side given saline assessed by cold sensation with alcohol soaked gauze.

SECONDARY OUTCOMES:
Difference in the percentage coverage of the incision (anterior-lateral approach) assessed by cold sensation | 1 hour post-block
  Difference in the percentage coverage of the incision (anterior-lateral approach) between the side given Ropivacaine versus the side given saline assessed by cold sensation with alcohol soaked gauze.
Difference in the percentage coverage of the incision (posterior approach) assessed by pin-prick | 1 hour post-block
  Difference in the percentage coverage of the incision (posterior approach) between the side given Ropivacaine versus the side given saline assessed by pin-prick (Von Frey filament).
Difference in the percentage coverage of the incision (anterior-lateral approach) assessed by pin-prick | 1 hour post-block
  Difference in the percentage coverage of the incision (anterior-lateral approach) between the side given Ropivacaine versus the side given saline assessed by pin-prick (Von Frey filament).
The percentage of participants with no sensory function (VAS = 0) assessed by Maximum pain during tonic heat stimulation test on the most superior part of the incision (posterior approach) | 1 hour post-block
  The percentage of patients with no sensory function (VAS = 0) assessed by Maximum pain during tonic heat stimulation test on the most superior part of the incision (posterior approach) on the side given Ropivacaine versus the side given saline.
The percentage of participants with no sensory function (VAS = 0) assessed by Maximum pain during tonic heat stimulation test on the most inferior part of the incision (posterior approach) | 1 hour post-block
  The percentage of patients with no sensory function (VAS = 0) assessed by Maximum pain during tonic heat stimulation test on the most inferior part of the incision (posterior approach) on the side given Ropivacaine versus the side given saline.
The percentage of participants with no sensory function (VAS = 0) assessed by Maximum pain during tonic heat stimulation test on the most superior part of the incision (anterior-lateral approach) | 1 hour post-block
  The percentage of patients with no sensory function (VAS = 0) assessed by Maximum pain during tonic heat stimulation test on the most superior part of the incision (anterior-lateral approach) on the side given Ropivacaine versus the side given saline.
The percentage of participants with no sensory function (VAS = 0) assessed by Maximum pain during tonic heat stimulation test on the most inferior part of the incision (anterior-lateral approach) | 1 hour post-block
  The percentage of patients with no sensory function (VAS = 0) assessed by Maximum pain during tonic heat stimulation test on the most inferior part of the incision (anterior-lateral approach) on the side given Ropivacaine versus the side given saline.
The percentage of participants with no sensory function (no pain detection) assessed by Heat pain detection threshold test on the most superior part of the incision (posterior approach) | 1 hour post-block
  The percentage of patients with no sensory function (no pain detection) assessed by Heat pain detection threshold test on the most superior part of the incision (posterior approach) on the side given Ropivacaine versus the side given saline.
The percentage of participants with no sensory function (no pain detection) assessed by Heat pain detection threshold test on the most inferior part of the incision (posterior approach) | 1 hour post-block
  The percentage of patients with no sensory function (no pain detection) assessed by Heat pain detection threshold test on the most inferior part of the incision (posterior approach) on the side given Ropivacaine versus the side given saline.
The percentage of participants with no sensory function assessed (no pain detection) by Heat pain detection threshold test on the most superior part of the incision (anterior-lateral approach) | 1 hour post-block
  The percentage of patients with no sensory function (no pain detection) assessed by Heat pain detection threshold test on the most superior part of the incision (anterior-lateral approach) on the side given Ropivacaine versus the side given saline.
The percentage of participants with no sensory function (no pain detection) assessed by Heat pain detection threshold test on the most inferior part of the incision (anterior-lateral approach) | 1 hour post-block
  The percentage of patients with no sensory function (no pain detection) assessed by Heat pain detection threshold test on the most inferior part of the incision (anterior-lateral approach) on the side given Ropivacaine versus the side given saline.
Estimation of the area with sensory loss assessed by cold sensation | 1 hour post-block
  Estimation of the area with sensory loss (including photo documentation) assessed by cold sensation (alcohol soaked gauze) on the side given Ropivacaine and the side given saline. Marked with the incisions.
Estimation of the area with sensory loss assessed by pin-prick | 1 hour post-block
  Estimation of the area with sensory loss (including photo documentation) assessed by pin-prick (Von Frey filament) on the side given Ropivacaine and the side given saline. Marked with the incisions.
The difference in MVIC (maximal voluntary isometric contraction) of the leg | 1 hour post-block
  The difference in MVIC (maximal voluntary isometric contraction) of the leg between the side given Ropivacaine versus the side given saline.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hägi-Pedersen, MD, PhD, Study Chair — Naestved Hospital; Kasper H Thybo, MD, Principal Investigator — Naestved Hospital
Locations (1):
- Zealand University Hospital, Køge, Køge, Køge, Denmark

IPD SHARING:
Plan to Share IPD: Yes
If data is requested by an editor it will be allowed

REFERENCES:
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Kehlet H, Dahl JB. Anaesthesia, surgery, and challenges in postoperative recovery. Lancet. 2003 Dec 6;362(9399):1921-8. doi: 10.1016/S0140-6736(03)14966-5. PMID 14667752
- [Background] Hojer Karlsen AP, Geisler A, Petersen PL, Mathiesen O, Dahl JB. Postoperative pain treatment after total hip arthroplasty: a systematic review. Pain. 2015 Jan;156(1):8-30. doi: 10.1016/j.pain.0000000000000003. PMID 25599296
- [Background] Fischer HB, Simanski CJ. A procedure-specific systematic review and consensus recommendations for analgesia after total hip replacement. Anaesthesia. 2005 Dec;60(12):1189-202. doi: 10.1111/j.1365-2044.2005.04382.x. PMID 16288617
- [Background] Thybo KH, Schmidt H, Hagi-Pedersen D. Effect of lateral femoral cutaneous nerve-block on pain after total hip arthroplasty: a randomised, blinded, placebo-controlled trial. BMC Anesthesiol. 2016 Mar 23;16:21. doi: 10.1186/s12871-016-0183-4. PMID 27006014
- [Background] Thybo KH, Mathiesen O, Dahl JB, Schmidt H, Hagi-Pedersen D. Lateral femoral cutaneous nerve block after total hip arthroplasty: a randomised trial. Acta Anaesthesiol Scand. 2016 Oct;60(9):1297-305. doi: 10.1111/aas.12764. Epub 2016 Jul 18. PMID 27426231
- [Background] Davies A, Crossley A, Harper M, O'Loughlin E. Lateral cutaneous femoral nerve blockade-limited skin incision coverage in hip arthroplasty. Anaesth Intensive Care. 2014 Sep;42(5):625-30. doi: 10.1177/0310057X1404200513. PMID 25233177